CLINICAL TRIAL: NCT04549467
Title: Efficacy of Dolutegravir Plus Lamivudine Compared to Dolutegravir Plus Tenofovir/Emtricitabine in HIV-1-infected Treatment-naïve Adults Without Baseline Genotyping Test (D2ARLING Study)
Brief Title: Efficacy of Dolutegravir Plus Lamivudine in HIV-1-infected Treatment-naïve Adults Without a Baseline Genotyping Test
Acronym: D2ARLING
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion IDEAA (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDEAA 002
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Hiv; HIV-1-infection
Keywords: hiv; antiretroviral treatment; dolutegravir; dual therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Lamivudine; dolutegravir; Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dolutegravir + lamivudine (Experimental): Dolutegravir 50 mg, 1 tablet QD plus lamivudine 300 mg, 1 tablet QD
  Interventions: Drug: Lamivudine 300 MG
- Dolutegravir + emtricitabine/tenofovir (FTC/TDF) (Active Comparator): Dolutegravir 50 mg, 1 tablet QD plus FTC/TDF 200/300 mg, 1 coformulated tablet QD
  Interventions: Drug: Emtricitabine / Tenofovir Disoproxil Pill

INTERVENTIONS:
Drug: Lamivudine 300 MG — Experimental arm
  Other Names: 3TC; dolutegravir
  Arms: Dolutegravir + lamivudine
Drug: Emtricitabine / Tenofovir Disoproxil Pill — Active Comparator
  Other Names: truvada; dolutegravir
  Arms: Dolutegravir + emtricitabine/tenofovir (FTC/TDF)

SUMMARY:
The purpose of this study is to evaluate the efficacy of DTG + 3TC versus DTG + TDF/FTC over 48 weeks in HIV-1 naive patients in a real life setting with no baseline HIV genotypic resistance testing available.

DETAILED DESCRIPTION:
This is a 48-week, Phase IV, randomized, open-label, to assess the non-inferior antiviral activity (VL < 50 c/ml) of 2DR DTG+3TC versus 3DR TDF/FTC + DTG over 48 weeks in HIV1 naïve adult patients without baseline GT available at Day 1 visit. Subjects will be stratified by screening HIV-1 RNA (≤100,000 c/mL or >100,000 c/mL) and Screening CD4+ cell count (≤ or >200 cells/mm3).

The study will comprise:

* a 28-day Screening Phase (which may be extended to 35 days to allow receipt of all Screening assessment results).
* an Open-label Randomized Phase (Day 1 to Week 48).

Approximately 200 HIV-1 naïve adult patients will be randomized 1:1 to receive 2DR DTG+3TC versus 3DR TDF/FTC + DTG for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject should be antiretroviral naïve (defined as <=10 days of prior therapy with any antiretroviral agent following a diagnosis of HIV 1 infection).
2. Age ≥ 18 years
3. Screening plasma HIV-1 RNA ≥1000 c/mL
4. CD4 cell count nadir: any value
5. Effective contraception for women of childbearing potential.
6. Informed consent form signed by patient and investigator

Exclusion Criteria:

1. History of suicide ideation, intention or action.
2. Evidence of HBV infection based on the results of testing at Screening* for HBV surface antigen (HBsAg), HBV core antibody (anti-HBc), HBV surface antibody (antiHBs or HBsAb), and HBV DNA as follows: Subjects positive for HBsAg are excluded; Subjects negative for anti-HBs and HBsAg but positive for anti-HBc and positive for HBV DNA are excluded.
3. Anticipated need for any HCV therapy during the first 48 weeks of the study.
4. Acute symptomatic HIV Infection.
5. Any active Opportunistic Infection (category C, CDC 2014).
6. Current pregnancy or breastfeeding.
7. No effective contraception for the women of childbearing.
8. Any verified Grade 4 laboratory abnormality. A single repeat test is allowed during the Screening period to verify a result.
9. ALT (Alanine Aminotransferase) ≥ 5 x upper limit of normal value (ULN) or AST (Aspartate Aminotransferase) ≥ 3 x ULN and bilirubinemia ≥ 1.5 x ULN (with 35% direct bilirubinemia).
10. Unstable liver disease (ascitis, encephalopathy, coagulopathy, hypoalbuminemia, oesophageal or gastric varices or persistent jaundice).
11. Creatinine clearance of <50 mL/min/1.73 m2 (Cockroft-Gault method).
12. History or presence of allergy to the trial drugs or their components.
13. Severe hepatic insufficiency (Child Pugh Class C).
14. Any available historical resistance test result.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Virologic Efficacy | 48 weeks
  To demonstrate the non-inferior antiviral activity (VL < 50 c/ml) of 2DR DTG+3TC versus 3DR TDF/FTC + DTG over 48 weeks in HIV-1 naïve adult patients without baseline genotypic resistance testing available. Endpoint: Proportion of subjects with plasma HIV-1 RNA <50 copies/mL (c/mL) at Week 48 using the FDA Snapshot algorithm [Missing, Switch or Discontinuation = Failure (MSD=F)] for the intent-to-treat exposed (ITT-E) population.

SECONDARY OUTCOMES:
Genetic barrier | 48 weeks
  To assess the selection / emergence of viral resistance in subjects meeting confirmed virologic withdrawal (CVW) criteria. Endpoint: incidence of treatment-emergent genotypic resistance to DTG and 3TC or TDF/FTC in subjects meeting CVW criteria.
Efficacy in presence of any major resistanceassociated mutation al baseline | 48 weeks
  To evaluate the antiviral activity of DTG + 3TC compared to DTG + TDF/FTC over time in patients with pre-existing viral resistance based on the presence of any major resistanceassociated mutation (IAS-USA 2019). Endpoint: Proportion of subjects with plasma HIV-1 RNA <50 copies/mL (c/mL) at Week 48 using the FDA Snapshot algorithm and The proportion of participants with HIV-1 RNA <50 or <200 copies/mL using the observed algorithm (excluding participants with missing data) in patients with pre-existing viral resistance based on the presence of any major resistance-associated mutation (IAS-USA 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Ezequiel Cordova, MD, Principal Investigator — Fundacion IDEAA
Locations (1):
- Fundacion IDEAA, Buenos Aires, Argentina

REFERENCES:
- [Derived] Cordova E, Hernandez Rendon J, Mingrone V, Martin P, Arevalo Calderon G, Seleme S, Ballivian J, Porteiro N. Efficacy of dolutegravir plus lamivudine in treatment-naive people living with HIV without baseline drug-resistance testing available (D2ARLING): 48-week results of a phase 4, randomised, open-label, non-inferiority trial. Lancet HIV. 2025 Feb;12(2):e95-e104. doi: 10.1016/S2352-3018(24)00294-7. Epub 2025 Jan 15. PMID 39826566
- See also: Fundacion IDEAA web page — http://fundacionideaa.com.ar/